CLINICAL TRIAL: NCT00707070
Title: Phase IV Study on Efficacy and Safety of the Combination Treatment Acitretin and Efalizumab in Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Combining Acitretin and Efalizumab in the Therapy of Chronic Plaque Psoriasis
Acronym: CobAcE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universita di Verona (Other)
Responsible Party: Giampiero Girolomoni, University of Verona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Gisondi 2; No grants were received
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2008-06-30 (Estimated); Status verified 2008-06

CONDITIONS: Chronic Plaque Psoriasis
Keywords: psoriasis; acitretin; efalizumab
MeSH Terms: conditions — Psoriasis | interventions — efalizumab; Acitretin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): efalizumab 1 mg/kg/week subcutaneous plus acitretin 0.4 mg/kg/day oral
  Interventions: Drug: efalizumab plus acitretin
- 2 (Placebo Comparator): efalizumab 1 mg/Kg/week subcutaneous plus oral placebo
  Interventions: Drug: efalizumab plus placebo

INTERVENTIONS:
Drug: efalizumab plus placebo — 1 mg/kg/week subcutaneous for 24 weeks
  Arms: 2
Drug: efalizumab plus acitretin — 1 mg/Kg/week for 24 weeks plus oral acitretin 0.4 mg/kg/day
  Arms: 1

SUMMARY:
It is a phase IV multicentric, placebo-controlled, clinical trial investigating the efficacy and safety of acitretin combined to efalizumab in the therapy of chronic plaque psoriasis. PASI 75 at week 24 will be the primary end point. PASI 75 at week 12, and PASI 50 at week 24 will be the secondary end points. Safety measures will be the monitoring of serum parameters including AST; ALT; gammaGT; creatinine; cholesterol and triglycerides.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18-70
* Women in postmenopausal
* Moderate to severe chronic plaque psoriasis in patients with contraindication, intolerance or non responsive to cyclosporine, methotrexate or PUVA
* PASI > 10 e/o BSA (Body Surface Area) > 10

Exclusion Criteria:

* Drug induced psoriasis
* Pustular or erythrodermic psoriasis
* Fertile women
* Pregnancy or lactation
* cholesterol > 230mg/dL e triglyceride > 200 mg/dL
* Known intolerance to efalizumab and acitretin
* Serious infection at enrollement
* History of previous neoplasia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-10 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
PASI 75 and PASI 50 at week 24 Physician Global Assessment | week 12 and 24

SECONDARY OUTCOMES:
SKINDEX 29 at week 24 and AST, ALT, cholesterol, triglycerides at week 12 and week 24 | week 24

CONTACTS AND LOCATIONS:
Overall Officials: Giampiero Girolomoni, Principal Investigator — Universita di Verona
Locations (1):
- Univeristy Hospital, Verona, Italy

REFERENCES:
- [Background] Gisondi P, Girolomoni G. Combination of efalizumab and acitretin in chronic plaque psoriasis. J Eur Acad Dermatol Venereol. 2008 Feb;22(2):247-8. doi: 10.1111/j.1468-3083.2007.02303.x. No abstract available. PMID 18211428